CLINICAL TRIAL: NCT07372521
Title: Measuring Small-Airways Disease Improvement After Step-up to Extrafine TRIple or High-dose ICS/LABA in Patients Uncontrolled on Medium Dose ICS/LABA eXploring T2 Inflammation: The MATRIX Real-life Observational Study
Brief Title: Measuring Small-Airways Disease Improvement After Step-up to Extrafine TRIple or High-dose ICS/LABA in Patients Uncontrolled on Medium Dose ICS/LABA eXploring T2 Inflammation
Acronym: MATRIX
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Ioannina (Other)
Collaborators: Attikon Hospital (Other); 424 General Military Hospital (Other); George Papanicolaou Hospital (Other); University Hospital of Patras (Other); University Hospital, Alexandroupolis (Other)
Responsible Party: Principal Investigator, Konstantinos Kostikas, Professor and Head Respiratory Medicine, University of Ioannina, Greece, University Hospital, Ioannina
Other Study IDs: RMDUoI-001; University Hospital Ioannina (Other: Respiratory Medicine Department, University of Ioannina, Greece)
Record Dates: First submitted 2026-01-11; First posted 2026-01-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma; Clinical Trials, Phase IV as Topic; Drug Therapy, Combination; LABA; LAMA; ICS; Oscillometry; Respiratory Function Tests; FeNO
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Males and females out-patients aged ≥18 years with uncontrolled asthma on ICS/LABA treatment

SUMMARY:
The goal of this observational study is to investigate the change in small airway function through the R5-R19 index in oscillometry at 12 weeks in adults with asthma.

The main question it aims to answer is: How can small airways dysfunction as evaluated by the oscillometry measure R5-19 be improved at 12 weeks, using 2 treatment arms (high-dose ICS regimen or medium dose efSITT)?

Researchers will compare the efficacy of either (1) high-dose ICS combinations (high-dose extrafine BDP/FF or high-dose efSITT BDP/FF/G) or (2) medium-dose efSITT (BDP/FF/G) to determine whether there is an improvement in small airways dysfunction and better asthma control in patients who are uncontrolled on medium-dose ICS/LABA.

Participants will take as drugs the Trimbow (BDP/FF/G) medium (100/6/10 μg) or high (200/6/10 μg) strengths or Foster (BDP/FF) high strength (200/6 μg); Visit the clinic three times with an one optional follow up visit, at the start (Visit 1: baseline), at 4 weeks (Visit 2), at 12 weeks (Visit 3) and the optional visit at 52 weeks (Visit 4).

DETAILED DESCRIPTION:
All data related to the study will be recorded for each participating patient by the investigator in a separate, specially designed Case Report Form (CRF) at the start of the study. The CRF pages are specifically designed to capture the information required by the study protocol, and the investigator will enter these data into the corresponding fields, ensuring consistency with the information documented in the patient's medical record.

All patients who sign the informed consent to participate in the study will be assigned a unique 5-digit identification number in the format of XX-XXX (first two digits represent the centre number and the last 3 digits the patient number), which will be recorded on all relevant study documents (CRF etc.). The patient's initials and full date of birth will not be recorded in the CRF to protect personal data, except in cases specifically permitted under the General Data Protection Regulation (GDPR).

• At all 3 Visits, the following assessments will be performed to all patients: (1) Evaluation of asthma control (ACT, ACQ-5), (2) Blood Eosinophil Counts (BEC, cells/mL and %), (3) FeNO (FeNO+, MGC Diagnostics, at 50 mL/sec and at 100 and 150 mL/sec to measure alveolar NO as a marker of SAD), (4) Forced Oscillometry Technique (FOT, Resmon PRO Full V3), measuring peripheral resistance (difference between resistance at 5Hz and 19Hz, R5-19), frequency resonance (Fres), area of reactance (AX), and reactance (X5), (5) Simple spirometry, including forced expiratory volume in 1 sec (FEV1), forced vital capacity (FVC), FEV1/FVC ratio, and forced expiratory flow at 25-75% of FVC (FEF25-75%), (6) Static lung volumes by body plethysmography, including total lung capacity (TLC), residual volume (RV), and functional residual capacity (FRC), (7) At the optional Visit 4 at 52 weeks, we will collect the previous parameters and the number of exacerbations (OCS courses, emergency department visits, hospitalizations).

eCRFs will be periodically reviewed by the principal investigator to minimize missing values. When NaN entries cannot be avoided, the amount, pattern, and assumed mechanism of missingness (missing completely at random, missing at random, or missing not at random) will be evaluated to determine the most appropriate statistical approach. Imputation methods may include mean or median imputation, random sample imputation, or multiple imputation, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Males and females out-patients aged ≥18 years providing written informed consent. [Note: Females are eligible if they are of non-childbearing potential or, if they are of childbearing potential, using or are willing to use appropriate contraceptive measures.]
* Physician-diagnosed asthma for at least 6 months
* Patients with uncontrolled asthma (ACT<20 or ACQ-5>1.5) on stable treatment with medium dose ICS/LABA for at least 12 weeks and with good adherence to treatment.
* Evidence of SAD as expressed by FEF25-75% <60% in spirometry.
* Ability to be trained to use properly a pMDI inhaler (with or without spacer as per physician's judgement).
* Documented decision in the patient's medical file for the (high-dose ICS regimen or medium dose efSITT) before the patient gets informed about his/her potential participation in the study.

Exclusion Criteria:

* Age <18 years
* Patients who have experienced a severe asthma exacerbation (i.e. receiving OCS for at least 3 days and/or antibiotics or need for hospitalisation) in the 4 weeks prior to the screening visit.
* Refusal or inability to give informed consent.
* Patients with COPD or other respiratory disease, e.g. bronchiectasis, cystic fibrosis, interstitial lung diseases or any other clinically or functionally significant lung disorder, cancer (except localized carcinomas), or other clinically significant comorbidities that may affect the outcomes measured.
* Long-term oxygen therapy at home.
* Pregnancy or lactation or planned pregnancy.
* Patients with a history of hypersensitivity or contraindications to any of the components of the study drug.
* Participation in interventional study within 30 days prior to enrolment or at least two half-life times of an investigational drug.
* Patient inability or incompliance to follow physician's instructions concerning treatment or study visits or unreliability, according to the physician evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with physician-diagnosed asthma, recruited from outpatient and/or inpatient clinics at participating hospitals.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Small airways function and Oscillometry | From January 2026 to June 2027
  Improvement in small airways function as evaluated by the oscillometry measure R5-19 (in cmH2O/L/s) at 12 weeks compared to baseline in the whole study population

SECONDARY OUTCOMES:
Pulmonary test function results and Questionnaires | From January 2026 to June 2027
  Change in R5-19 (cmH2O/L/s, at 4 weeks), Change in FEF25-75% (% pred., at 4 and 12 weeks), Change in FEV1 (L, at 4 and 12 weeks), Change in residual volume (RV) (% pred., at 4 and 12 weeks), Change in total lung capacity (TLC) (% pred., at 4 and 12 weeks), Change in FeNO (ppb, at 4 and 12 weeks), Change in asthma control test (ACT) (at 4 and 12 weeks), Change in asthma quality of life (mini-AQLQ) (at 4 and 12 weeks)

OTHER OUTCOMES:
Optional evaluation (at 52 weeks) | From January 2026 to June 2027
  Change in R5-19 (at 4 weeks), Change in FEF25-75% (at 4 and 12 weeks), Change in FEV1 (at 4 and 12 weeks), Change in residual volume (RV) (at 4 and 12 weeks), Change in total lung capacity (TLC) (at 4 and 12 weeks), Change in FeNO (at 4 and 12 weeks), Change in asthma control test (ACT) (at 4 and 12 weeks), Change in asthma quality of life (mini-AQLQ) (at 4 and 12 weeks) Exacerbations (OCS courses, emergency department visits, hospitalizations) in the follow-up period and comparison to the exacerbation history in the previous year

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting after the date of publication.
Access Criteria: Individual participant data (IPD) and supporting information from this trial will be freely available to qualified researchers following the publication of the trial results. Access will include the de-identified participant-level dataset, study protocol, and statistical analysis plan. Researchers may request the data through the corresponding data repository link.

REFERENCES:
- [Background] Gogali A, Kostikas K, Kyriakopoulos C, Potonos D, Porpodis K, Tsiouprou I, Fouka E, Tryfon S, Papadopoulou E, Kipourou M, Katsoulis K. Managing Small Airways Dysfunction in COPD Patients in Real Life Under Fixed Triple Combination of Beclomethasone/Formoterol/Glycopyrronium: The MASCOT Real World Evidence Study. Int J Chron Obstruct Pulmon Dis. 2025 May 23;20:1651-1663. doi: 10.2147/COPD.S513350. eCollection 2025. PMID 40433397
- [Background] Bhakta NR, McGowan A, Ramsey KA, Borg B, Kivastik J, Knight SL, Sylvester K, Burgos F, Swenson ER, McCarthy K, Cooper BG, Garcia-Rio F, Skloot G, McCormack M, Mottram C, Irvin CG, Steenbruggen I, Coates AL, Kaminsky DA. European Respiratory Society/American Thoracic Society technical statement: standardisation of the measurement of lung volumes, 2023 update. Eur Respir J. 2023 Oct 12;62(4):2201519. doi: 10.1183/13993003.01519-2022. Print 2023 Oct. PMID 37500112
- [Background] Santanello NC, Zhang J, Seidenberg B, Reiss TF, Barber BL. What are minimal important changes for asthma measures in a clinical trial? Eur Respir J. 1999 Jul;14(1):23-7. doi: 10.1034/j.1399-3003.1999.14a06.x. PMID 10489824
- [Background] Stanojevic S, Kaminsky DA, Miller MR, Thompson B, Aliverti A, Barjaktarevic I, Cooper BG, Culver B, Derom E, Hall GL, Hallstrand TS, Leuppi JD, MacIntyre N, McCormack M, Rosenfeld M, Swenson ER. ERS/ATS technical standard on interpretive strategies for routine lung function tests. Eur Respir J. 2022 Jul 13;60(1):2101499. doi: 10.1183/13993003.01499-2021. Print 2022 Jul. PMID 34949706
- [Background] Juniper EF, Buist AS, Cox FM, Ferrie PJ, King DR. Validation of a standardized version of the Asthma Quality of Life Questionnaire. Chest. 1999 May;115(5):1265-70. doi: 10.1378/chest.115.5.1265. PMID 10334138
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Galant SP, Kuks PJM, Kole TM, Kraft M, Siddiqui S, Fabbri LM, Beghe B, Rabe KF, Papi A, Brightling CE, Singh D, Kocks JWH, Franzini L, Vonk JM, Kerstjens HAM, Heijink IH, Pouwels SD, Slebos DJ, van den Berge M. Assessment of the role of small airway dysfunction in relation to exacerbation risk in patients with well controlled asthma (ATLANTIS): an observational study. Lancet Respir Med. 2025 Nov;13(11):990-1000. doi: 10.1016/S2213-2600(25)00283-8. Epub 2025 Sep 29. PMID 41038213
- [Background] 2025 GINA Strategy Report [Internet]. Global Initiative for Asthma - GINA 2025 [cited 2025 Oct 28]. Available from: https://ginasthma.org/2025-gina-strategy-report/).
- [Background] Papi A, Singh D, Virchow JC, Canonica GW, Vele A, Georges G. Normalisation of airflow limitation in asthma: Post-hoc analyses of TRIMARAN and TRIGGER. Clin Transl Allergy. 2022 Apr 17;12(4):e12145. doi: 10.1002/clt2.12145. eCollection 2022 Apr. PMID 35450196
- [Background] Quaranta VN, Montagnolo F, Portacci A, Dragonieri S, Granito M, Rociola G, Ferrulli S, Maselli L, Carpagnano GE. Steady Quiet Asthma Without Biologics: One-Year Outcomes of Single-Inhaler Triple Therapy for Severe Asthma with Small Airway Dysfunction. J Clin Med. 2025 Aug 7;14(15):5602. doi: 10.3390/jcm14155602. PMID 40807224
- [Background] Carpagnano GE, Scioscia G, Lacedonia D, Stornelli SR, Irene Quarato CM, Soccio P, Resta O, Foschino Barbaro MP. Treatment response according to small airways disease status: The effects of high-strength extrafine pMDI beclomethasone dipropionate/formoterol fumarate in fixed dose combination in moderate uncontrolled asthmatic patients. Pulm Pharmacol Ther. 2020 Feb;60:101879. doi: 10.1016/j.pupt.2019.101879. Epub 2019 Dec 20. PMID 31866498
- [Background] Scichilone N, Battaglia S, Sorino C, Paglino G, Martino L, Paterno A, Santagata R, Spatafora M, Nicolini G, Bellia V. Effects of extra-fine inhaled beclomethasone/formoterol on both large and small airways in asthma. Allergy. 2010 Jul;65(7):897-902. doi: 10.1111/j.1398-9995.2009.02306.x. Epub 2010 Jan 28. PMID 20121764
- [Background] Virchow JC, Kuna P, Paggiaro P, Papi A, Singh D, Corre S, Zuccaro F, Vele A, Kots M, Georges G, Petruzzelli S, Canonica GW. Single inhaler extrafine triple therapy in uncontrolled asthma (TRIMARAN and TRIGGER): two double-blind, parallel-group, randomised, controlled phase 3 trials. Lancet. 2019 Nov 9;394(10210):1737-1749. doi: 10.1016/S0140-6736(19)32215-9. Epub 2019 Sep 30. PMID 31582314
- [Background] Kraft M, Richardson M, Hallmark B, Billheimer D, Van den Berge M, Fabbri LM, Van der Molen T, Nicolini G, Papi A, Rabe KF, Singh D, Brightling C, Siddiqui S; ATLANTIS study group. The role of small airway dysfunction in asthma control and exacerbations: a longitudinal, observational analysis using data from the ATLANTIS study. Lancet Respir Med. 2022 Jul;10(7):661-668. doi: 10.1016/S2213-2600(21)00536-1. Epub 2022 Mar 2. PMID 35247313
- [Background] Postma DS, Brightling C, Baldi S, Van den Berge M, Fabbri LM, Gagnatelli A, Papi A, Van der Molen T, Rabe KF, Siddiqui S, Singh D, Nicolini G, Kraft M; ATLANTIS study group. Exploring the relevance and extent of small airways dysfunction in asthma (ATLANTIS): baseline data from a prospective cohort study. Lancet Respir Med. 2019 May;7(5):402-416. doi: 10.1016/S2213-2600(19)30049-9. Epub 2019 Mar 12. PMID 30876830